CLINICAL TRIAL: NCT05518110
Title: PaTcH Trial: A Phase 2 Study to Explore Primary and Emerging Resistance Mechanisms in Patients With Metastatic Refractory Pancreatic Cancer Treated With Trametinib and Hydroxychloroquine
Brief Title: PaTcH Study: A Phase 2 Study of Trametinib and Hydroxychloroquine in Patients With Metastatic Refractory Pancreatic Cancer
Acronym: PaTcH
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Trials Ireland (Network)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTRIAL-IE 20-27; 2021-006276-16 (EudraCT Number)
Record Dates: First submitted 2022-07-22; First posted 2022-08-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Pancreatic Cancer
Keywords: Metastatic refractory; Primary and emerging resistance mechanisms
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — trametinib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- PaTcH (Experimental): All eligible patients will be treated with trametinib 2mg and hydroxychloroquine 1200mg daily (600mg twice a day (BID)) orally. Treatment will be continuous in treatment cycles lasting 28 days, and will continue until radiological or clinical progression of disease, unacceptable toxicity or consent withdrawal.
  Interventions: Drug: Trametinib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Trametinib — 2mg of Trametinib (orally) daily.
Drug: Hydroxychloroquine — 1200mg of Hydroxychloroquine (orally; 600mg twice a day (BID)) daily.

SUMMARY:
This study is designed to investigate the means by which cancer resists treatment can be overcome by a combination of an established anticancer drug, trametinib, with hydroxychloroquine.

DETAILED DESCRIPTION:
The study is a multi-centre single arm Phase 2 clinical trial to explore primary and emerging resistance mechanisms in patients with metastatic refractory pancreatic cancer treated with trametinib and hydroxychloroquine. This study will include 10-22 patients with metastatic pancreatic cancer who have previously progressed on at least one line of systemic therapy.

ELIGIBILITY:
Inclusion Criteria:

Each patient must meet all of the following inclusion criteria to be eligible for the study:

1. Patients must have pathologically confirmed advanced metastatic pancreatic adenocarcinoma or poorly differentiated pancreatic adenocarcinoma that is amenable to tumour biopsy.
2. Patients have received at least one line of systemic therapy for metastatic disease and not be amenable to surgical resection.
3. Patients must have measurable disease by RECIST 1.1 criteria.
4. Age ≥18 years.
5. ECOG performance status ≤ 1
6. Patients must have normal organ and marrow function as defined below:

   1. Serum creatinine ≤ 1.5 x ULN.
   2. Adequate hepatic function defined by:

      * total bilirubin level ≤ 1.5 × ULN,
      * an AST, level ≤ 2.5 × ULN, and an ALT level ≤ 2.5 × ULN (or, for subjects with documented metastatic disease to the liver, AST and ALT levels ≤ 5 × ULN)
   3. Hematological eligibility parameters:

      * Absolute Neutrophil count ≥ 1.5 x 109/L
      * Platelet count ≥100 x109/L
      * Hemoglobin ≥ 9 g/dL
7. Ability of subject to understand and the willingness to sign a written informed consent document.
8. Women of child-bearing potential or sexually active males must agree to use highly effective contraceptive measures. This applies from starting treatment until at least 16 weeks after the last study drug administration. The investigator or a designated associate is required to advise the patient how to achieve an adequate birth control. Highly effective contraception is defined in the study as methods that achieve a failure rate of less than 1% per year when used consistently and correctly. Such methods include:

I. Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal). II. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable and implantable). III. Intrauterine device (IUD). IV. Intrauterine hormone-releasing system (IUS). V. Bilateral tubal occlusion. VI. Successfully vasectomised partner. VII. Sexual abstinence.

Exclusion Criteria:

Patients are excluded from the study if any of the following exclusion criteria apply:

1. Persisting toxicity related to prior therapy (CTCAE Grade > 1); however alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤2 AEs not constituting a safety risk based on investigator's judgment are acceptable.
2. Prior treatment with a MEK inhibitor
3. Known history of testing positive for Human Immunodeficiency Virus (HIV) or known acquired immunodeficiency syndrome.
4. Any significant disease that, in the opinion of the investigator, may impair the patient's tolerance of study treatment.
5. Patients who are receiving any other investigational agents within 28 days before start of study treatment.
6. Prior organ transplantation including allogenic stem-cell transplantation.
7. Patients with known central nervous system metastases.
8. Active uncontrolled infection, requiring systemic therapy.
9. Clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (≥ New York Heart Association Classification Class II), or serious cardiac arrhythmia requiring medication.
10. Severe left ventricular dysfunction as defined by ejection fraction < 45%
11. Other severe acute or chronic medical conditions including colitis, inflammatory bowel disease, pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behaviour; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
12. Known maculopathy of the eye
13. Known history or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
14. Screening corrected QT interval by Fridericia (QTcF) > 500 msec
15. Pregnant women and breastfeeding mothers are excluded due to unknown impact on embryos or infants
16. Known prior severe hypersensitivity to investigational products or any component in its formulation.
17. Concurrent use of medicines known to induce retinal toxicity (e.g. tamoxifen) or QT interval prolonging agents.
18. Known congenital or documented acquired QT prolongation.
19. Uncorrected hypokalemia and/or hypomagnesemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Patients free of disease progression | Twelve weeks from starting treatment.
  The percentage of patients free of disease progression at 12 weeks from starting treatment into the study as determined by radiographic disease assessments per RECIST version 1.1.

SECONDARY OUTCOMES:
Tumour Response Rate | Twelve weeks following the 15th and 22nd patients.
  Confirmed tumour response rate as assessed by RECIST version 1.1.
Duration of Response | Through study treatment, an average of 1 year
  Confirmed duration of response as assessed by RECIST version 1.1.
Overall Survival | Through study completion, an average of five years
  Overall Survival
Safety and tolerability | Through study treatment, an average of one year
  The safety and tolerability of this regimen as measured by incidence of adverse events reported and toxicity evaluation as per the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.

OTHER OUTCOMES:
The number of successfully established organoid cultures per patient before and on treatment | Through study treatment, an average of one year
  The number of successfully established organoid cultures per patient from biopsies of patients with pancreatic cancer being treated with trametinib and hydroxychloroquine before treatment and on treatment.
Organoid resistance to trametinib and hydroxychloroquine | Through study treatment, an average of one year
  The number of organoids resistant to trametinib and hydroxychloroquine treatment as measured by proliferation and apoptosis rates.
Resistance mechanisms and their potential therapies in vitro | Through study treatment, an average of one year
  A list of potential resistance mechanisms and their potential therapies that can be tested on in vitro organoid cultures.
Comparison of new methods of multi-omics data integration vs existing models using AUROC | Through study treatment, an average of one year
  A comparison the performance of new methods of multi-omics data integration against existing models using AUROC (area under the receiver operating characteristic) analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Austin Duffy, Principal Investigator — Mater Misericordiae University Hospital
Locations (2):
- Ireland (2):
  - Mater Misericordiae University Hospital, Dublin
  - St Vincent's University Hospital, Dublin

IPD SHARING:
Plan to Share IPD: Yes
Pseudo-anonymised biological samples will be shared with the University College of Dublin for performance of the translational sub-study throughout the study.
Supporting Information: Study Protocol, ICF
Time Frame: Study duration
Access Criteria: IPD data will be shared for all patients who provide informed consent to participation in the sub-study.